CLINICAL TRIAL: NCT02689388
Title: The Use of Post-operative Regional Analgesia Rather Than Systemic Analgesia to Decrease the Incidence of Post-operative Delirium After Acute Hip Fracture Surgery? A Prospective Randomized-controlled Double-blinded Pilot Study.
Brief Title: Evaluating the Addition of Regional Analgesia to Reduce Postoperative Delirium in Patients Having Hip Fracture Surgery.
Acronym: RASAPOD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility
Sponsor: Auckland City Hospital (Other Government)
Responsible Party: Principal Investigator, Assoc. Prof Timothy Short, Consultant Anesthetist, Auckland City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ADHB_6925
Record Dates: First submitted 2016-02-18; First posted 2016-02-24 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Delirium; Hip Fracture
Keywords: analgesia; regional analgesia; femoral nerve block; older persons; frail
MeSH Terms: conditions — Delirium; Hip Fractures; Agnosia | interventions — Nerve Block; Anesthesia, Conduction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Anesthesia with nerve block (Active Comparator): Femoral Nerve Block
  Interventions: Procedure: Femoral Nerve Block
- General Anesthesia no nerve block (No Intervention): No femoral Nerve Block

INTERVENTIONS:
Procedure: Femoral Nerve Block — Use of femoral nerve block as part of general anesthesia
  Other Names: Nerve Block; Regional Anesthesia
  Arms: General Anesthesia with nerve block

SUMMARY:
Post operative delirium is common after hip fracture surgery and is associated with increased length of hospital stay, delayed recovery and increased mortality. Postoperative delirium can also decrease a patient's quality of life and increase treatment costs. Anesthesia and pain relief (analgesia) treatments may also influence the incidence of delirium, but more research is needed into which techniques are effective in improving patient outcomes, care and decreasing costs. This pilot study compares the addition of regional analgesia as part of general anesthesia to determine the incidence of delirium following hip surgery. This is a collaborative study involving anesthesia, orthopedic surgery and geriatrics in the improvement of patient care.

ELIGIBILITY:
Inclusion criteria (must meet all 3):

* Greater than or equal to 65 years
* Have a hip fracture requiring surgery
* Written informed consent for participation of study prior to surgery.

Exclusion criteria:

* Contraindication to peripheral nerve block or local anaesthetics
* Unable to do delirium or cognitive testing due to language, vision or hearing impairment
* Unable to communicate with research staff due to language barriers
* History of chronic opioid use (longer than 1 month)
* Contraindication to general anesthesia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08-28 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The incidence of post-operative delirium after hip fracture surgery | immeidately to 5 days post operatively
  Identify the our local incidence of post operative delirium diagnosed with 3D-CAM (3 Minute Diagnostic Assessment for Confusion Assessment Method)

SECONDARY OUTCOMES:
Decreased recovery time after surgery | immediately - immediately - 90 days
  reduction in length of stay and recovery time
Decrease post-operative opioid consumption | immediately - immediately - 90 days
  reduction in the requirement for systemic/opiod analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Tin L Chiu, MBChB, Principal Investigator — Auckland City Hospital - Anaesthesia and Peri-Operative Medicine
Locations (1):
- Auckland City Hopsital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share individual subject data

REFERENCES:
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043